CLINICAL TRIAL: NCT02808143
Title: A Phase 1 Dose-Escalation Study of Intravesical MK-3475 and Bacillus Calmette-Guerin (BCG) in Subjects With High Risk and BCG-Refractory Non-Muscle-Invasive Bladder Cancer
Brief Title: Pembrolizumab and BCG Solution in Treating Patients With Recurrent Non-Muscle-Invasive Bladder Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Joshua Meeks, Joshua Meeks, MD, PhD, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 15U06; STU00202754 (CTRP (Clinical Trial Reporting Program)); NU 15U06 (Other: Northwestern University); P30CA060553 (NIH); NCI-2016-00664 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-05-25; First posted 2016-06-21 (Estimated); Results first posted 2022-10-20 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Recurrent Bladder Carcinoma; Stage 0a Bladder Urothelial Carcinoma; Stage 0is Bladder Urothelial Carcinoma; Stage I Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, BCG solution) (Experimental): PRE-INDUCTION PHASE: Patients receive pembrolizumab intravesically once on day -14.
  INDUCTION PHASE: Patients receive BCG solution intravesically once weekly for 6 weeks at weeks 0-5 and pembrolizumab intravesically every 2 weeks at weeks 0, 2, and 4.
  MAINTENANCE PHASE: Beginning 2 weeks after the last dose of BCG solution, patients receive pembrolizumab intravesically every 2 weeks for 12 weeks at weeks 7, 9, 11, 13, 15, and 17 for a total of 6 doses. Patients then receive pembrolizumab intravesically every 4 weeks at weeks 21, 25, 29, 33, 37, 41, 45, and 49 for a total of 8 doses.
  Interventions: Biological: BCG Solution; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Pharmacological Study

INTERVENTIONS:
Biological: BCG Solution — Given intravesically
  Other Names: Bacillus Calmette-Guerin Solution; TICE BCG Solution
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given intravesically
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Pharmacological Study — Correlative studies

SUMMARY:
The purpose of this study is to evaluate the efficacy (the effect of drug on tumor) and the tolerability (the effect of drug on the body) of pembrolizumab, when given as a single agent in patients with bladder tumors. Another purpose of the study is to see what tumor characteristics are associated with increased efficacy of the pembrolizumab. Pembrolizumab (MK-3475) is an antibody (a human protein that sticks to a part of the tumor and/or immune cells) designed to allow the body's immune system to work against tumor cells. Pembrolizumab is Food and drug Administration (FDA) approved for the treatment of advanced melanoma (a type of skin cancer) and some types of lung cancer. It is not yet approved by the United States Food and Drug Administration (USFDA) for bladder cancer, hence it is considered an investigational agent for this disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of the study drug (pembrolizumab [MK-3475]) when administered intravesically in combination with BCG in patients with high risk or BCG-refractory non-muscle-invasive bladder cancer (up to the individual maximum tolerated dose of each drug alone).

SECONDARY OBJECTIVES:

I. To describe the dose limiting toxicities (DLTs) of MK-3475 in combination with BCG in this population.

II. To assess the safety and tolerability of the combination of MK-3475 and BCG in subjects with high risk or BCG-refractory non-muscle-invasive bladder cancer.

TERTIARY OBJECTIVES:

I. To characterize the pharmacokinetics (PK) of MK-3475 in both blood and urine when administered intravesically in combination with BCG.

II. To measure humoral and cellular responses to tumor antigens on serum and urine samples by measuring the levels of cytokines (ie, interleukin [IL]-2, IL-6, IL-8, IL-10, IL-18, interferon gamma [IFN-gamma] and tumor necrosis factor alpha [TNF-alpha]) and peripheral blood lymphocyte phenotype throughout treatment.

III. To determine the response rate in terms of complete pathologic response in this population assessed when patient undergoes cystoscopies (weeks 17, 25, 33, 41, and 49 if applicable).

IV. To document the progression rate associated with the combination of intravesical MK-3475 and BCG in patients with high risk or BCG-refractory non-muscle-invasive bladder cancer.

V. To evaluate the relationship between tumor biomarkers programmed cell death (PD)-ligand (L)1, PD-L2, PD-1 as defined by immunohistochemistry (IHC) and adverse effects and recurrence rate.

OUTLINE: This is a dose-escalation study of pembrolizumab.

PRE-INDUCTION PHASE: Patients receive pembrolizumab intravesically once on day -14.

INDUCTION PHASE: Patients receive BCG solution intravesically once weekly for 6 weeks at weeks 0-5 and pembrolizumab intravesically every 2 weeks at weeks 0, 2, and 4.

MAINTENANCE PHASE: Beginning 2 weeks after the last dose of BCG solution, patients receive pembrolizumab intravesically every 2 weeks for 12 weeks at weeks 7, 9, 11, 13, 15, and 17 for a total of 6 doses. Patients then receive pembrolizumab intravesically every 4 weeks at weeks 21, 25, 29, 33, 37, 41, 45, and 49 for a total of 8 doses.

After completion of study treatment, patients are followed up every 3 months for 2 years, every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically documented recurrence of non-muscle-invasive bladder carcinoma (T1HG, T1HG after repeat transurethral resection [reTUR]) or BCG refractory; if patient has received BCG they can be Ta, Tis, or T1)
* Patients must have persistent high grade disease OR be BCG refractory, defined as either:

  * Recurrence within 6 months of receiving at least 2 courses of intravesical BCG (at least 5 or 6 inductions and at least 2 or 3 maintenance doses) or
  * T1 high grade disease at the first evaluation following induction BCG alone (at least 5 of 6 induction doses)
* Patients must agree to provide tissue from archival biopsy samples or newly obtained excisional biopsy of a tumor lesion

  * NOTE: Patients who do not have available specimens from previous biopsy or do not agree to provide this tissue are not eligible; cytological specimens will not be acceptable; availability of tissue must be confirmed at the time of registration, but the actual sample does not have to be received in order to complete registration
* Patients must have received one course of induction treatment with BCG (4-6 weekly doses), irrespective of the interval since last treatment; patients are allowed to have received any number of prior chemotherapy instillations

  * NOTE: Patients may have received prior intravesical interferon
* All patients must have imaging (computed tomography [CT] scan or magnetic resonance imaging [MRI]) documenting normal upper urinary tracts and absence of locally advanced bladder cancer within 60 days prior to study registration
* Have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Absolute neutrophil count (ANC) >= 1,500 /mcL within 14 days prior to registration
* Platelets >= 100,000 / mcL within 14 days prior to registration
* Hemoglobin >= 9 g/dL or >= 5.6 mmol/L within 14 days prior to registration
* Serum creatinine =< 1.5 X upper limit of normal (ULN) OR measured or calculated (creatinine clearance should be calculated per institutional standard) creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 60 mL/min for subject with creatinine levels > 1.5 X institutional ULN within 14 days prior to registration
* Serum total bilirubin =< 1.5 X ULN OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN within 14 days prior to registration
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 X ULN within 14 days prior to registration
* International normalized ratio (INR) or prothrombin time (PT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within therapeutic range of intended use of anticoagulants within 14 days prior to registration
* Activated PTT (aPTT) =< 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants within 14 days prior to registration
* Females of child-bearing potential (FOCBP) and males must agree to use adequate contraception (e.g. hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 120 days following completion of therapy; should a female patient become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately;

  * NOTE: A FOCBP is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria
  * Has not undergone a hysterectomy or bilateral oophorectomy
  * Has had menses at any time in the preceding 12 consecutive months (and therefore has not been naturally postmenopausal for > 12 months)
* FOCBP must have a negative urine or serum pregnancy test within 7 days prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Patients must have the ability to understand and the willingness to sign a written informed consent prior to registration on study

Exclusion Criteria:

* Patients who have had chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day -14 or who have not recovered (to =< grade 1 or baseline) from adverse events due to a previously administered agent are not eligible

  * Note: subjects with =< grade 2 neuropathy are an exception to this criterion and do qualify for the study
  * Note: if subject received major surgery within 4 weeks prior to day -14, they must have recovered adequately from the toxicity and/or complications per PI discretion
* Patients may not be receiving any other investigational agents within 4 weeks of the first dose of treatment
* Patients who have received a prior monoclonal antibody within 4 weeks prior to study day -14 or who have not recovered (to =< grade 1 or baseline) from adverse events due to agents administered more than 4 weeks earlier are not eligible
* Patients who have a diagnosis of immunodeficiency (per PI discretion) or who have received treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF agents within 2 weeks prior to study registration are not eligible

  * NOTE: patients who have received acute, low-dose, systemic immunosuppressant medications (eg, one-time dose of dexamethasone for nausea) may be enrolled in the study; the use of inhaled corticosteroids and mineralocorticoids (eg, fludrocortisone) is allowed
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475 are not eligible AND/OR patients who have had prior exposure to compounds of similar chemical or biologic composition to MK-3475 are not eligible
* Patients who have documentation of an uncontrolled intercurrent illness (as noted in their medical records) including, but not limited to any of the following, are not eligible

  * Ongoing or active infection requiring systemic treatment
  * Symptomatic congestive heart failure (New York Heart Association cardiac disease class III or IV)
  * Unstable angina pectoris
  * Myocardial infarction within the previous 3 months
  * Unstable cardiac arrhythmias
  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Any other illness or condition that the treating investigator feels would interfere with study compliance or would compromise the patient's safety or study endpoints
* Female patients who are pregnant or nursing are not eligible
* Patients who have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to BCG are not eligible
* Patients who have had an active infection requiring systemic therapy within 1 week prior to day -14 are not eligible UNLESS they are symptom-free and have a negative culture at the time of dosing on day -14
* Patients who received a live, attenuated vaccine within 4 weeks before study registration or are anticipated to require such a live attenuated vaccine are not eligible; NOTE: Influenza vaccination should be given during influenza season only (approximately October to March); patients must not receive live, attenuated influenza vaccine (e.g., FluMist) within 4 weeks prior to study registration or at any time during the study
* Patients who are known to be (i.e. documented in medical records) human immunodeficiency virus (HIV) positive are not eligible
* Patients with active tuberculosis are not eligible
* Patients with known active hepatitis B (chronic or acute; defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C are not eligible

  * NOTE: patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible; HBV deoxyribonucleic acid (DNA) must be obtained in these patients 14 days prior to study registration
  * NOTE: patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA)
* Patients who have a history of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins are not eligible
* Patients with an active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs); replacement therapy (eg. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Patients with a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; subjects with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; subjects with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Patients with history of interstitial lung disease or active, non-infectious pneumonitis are not eligible

  * NOTE: history of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Treatment with systemic immunostimulatory agents (including but not limited to IFNs, IL-2) within 6 weeks or five half-lives of the drug, whichever is shorter, prior to study registration are not eligible
* Patients who received prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways) are not eligible
* Patients who have a history of prior malignancy are not eligible; please NOTE the following exceptions when patient has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy

  * Basal cell carcinoma of the skin
  * Squamous cell carcinoma of the skin
  * In situ cervical cancer
* Patients who have a history of an allogeneic tissue/solid organ transplant are not eligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-02-10 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Meeks, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Derived] Meghani K, Cooley LF, Choy B, Kocherginsky M, Swaminathan S, Munir SS, Svatek RS, Kuzel T, Meeks JJ. First-in-human Intravesical Delivery of Pembrolizumab Identifies Immune Activation in Bladder Cancer Unresponsive to Bacillus Calmette-Guerin. Eur Urol. 2022 Dec;82(6):602-610. doi: 10.1016/j.eururo.2022.08.004. Epub 2022 Aug 23. PMID 36008193

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC); Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BCG): PRE-INDUCTION PHASE: Patients receive pembrolizumab intravesically once on day -14.
  INDUCTION PHASE: Patients receive BCG solution intravesically once weekly for 6 weeks at weeks 0-5 and pembrolizumab intravesically every 2 weeks at weeks 0, 2, and 4.
  MAINTENANCE PHASE: Beginning 2 weeks after the last dose of BCG solution, patients receive pembrolizumab intravesically every 2 weeks for 12 weeks at weeks 7, 9, 11, 13, 15, and 17 for a total of 6 doses. Patients then receive pembrolizumab intravesically every 4 weeks at weeks 21, 25, 29, 33, 37, 41, 45, and 49 for a total of 8 doses.
  BCG Solution: Given intravesically
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given intravesically
  Pharmacological Study: Correlative studies
Period: Pre-Induction Period
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BCG)
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0
Period: Induction Period
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BCG)
Started | 3 | 6
Completed | 3 | 6
Not Completed | 0 | 0
Period: Maintenance Phase
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BCG)
Started | 3 | 6
Completed | 1 | 1
Not Completed | 2 | 5
Not completed — Disease recurrence | 1 | 3
Not completed — Disease progression | 1 | 2
Period: Survival Follow-Up
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BCG)
Started (Once off treatment, patients were followed clinically for disease recurrence and survival according to protocol schedule until death, withdrawal, or end of study (whichever occurs first).) | 3 | 6
Completed | 0 | 0
Not Completed | 3 | 6
Not completed — Still in survival Follow-up | 2 | 3
Not completed — Disease recurrence | 0 | 2
Not completed — Adverse Event | 0 | 1
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC): PRE-INDUCTION PHASE: Patients receive pembrolizumab intravesically once on day -14.
  INDUCTION PHASE: Patients receive BCG solution intravesically once weekly for 6 weeks at weeks 0-5 and pembrolizumab intravesically every 2 weeks at weeks 0, 2, and 4.
  MAINTENANCE PHASE: Beginning 2 weeks after the last dose of BCG solution, patients receive pembrolizumab intravesically every 2 weeks for 12 weeks at weeks 7, 9, 11, 13, 15, and 17 for a total of 6 doses. Patients then receive pembrolizumab intravesically every 4 weeks at weeks 21, 25, 29, 33, 37, 41, 45, and 49 for a total of 8 doses.
  BCG Solution: Given intravesically
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given intravesically
  Pharmacological Study: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC) | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 3 | 6 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 5 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 8
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 2 | 4 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Cancer Stage at Baseline [Count of Participants; unit: Participants] — The TNM staging system is the common language in which oncology health professionals can communicate on the cancer extent for individual patients as a basis for decision making on treatment management and individual prognosis but can also be used, to inform and evaluate treatment guidelines. Tumors confined to the mucosa and invading the lamina propria are classified as stage Ta and T1, respectively, according to the Tumour, Node, Metastasis (TNM) classification system. Intra-epithelial, high-grade (HG) tumors confined to the mucosa are classified as CIS (Tis).
  Participants
    TaHG | 0 | 2 | 2
    TaHG + CIS | 1 | 1 | 2
    Tis | 1 | 2 | 3
    T1 | 1 | 0 | 1
    T1HG | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Determine the MTD of the study drug (MK-3475) when administered intravesically in combination with BCG in patients with high risk or BCG-refractory non-muscle-invasive bladder cancer (up to the individual maximum tolerated dose of each drug alone). The MTD will be defined as the highest dose that causes dose limiting toxicities (DLTs) in <2 of 6 patients graded by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: Up to 9 weeks
Measure: Number; unit: mg/kg Pembrolizumab
Groups:
- Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) & Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC): PRE-INDUCTION PHASE: Patients receive pembrolizumab intravesically once on day -14.
  INDUCTION PHASE: Patients receive BCG solution intravesically once weekly for 6 weeks at weeks 0-5 and pembrolizumab intravesically every 2 weeks at weeks 0, 2, and 4.
  MAINTENANCE PHASE: Beginning 2 weeks after the last dose of BCG solution, patients receive pembrolizumab intravesically every 2 weeks for 12 weeks at weeks 7, 9, 11, 13, 15, and 17 for a total of 6 doses. Patients then receive pembrolizumab intravesically every 4 weeks at weeks 21, 25, 29, 33, 37, 41, 45, and 49 for a total of 8 doses.
  BCG Solution: Given intravesically Laboratory Biomarker Analysis: Correlative studies Pembrolizumab: Given intravesically Pharmacological Study: Correlative studies
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) & Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC)
Number analyzed (Participants) | 9
mg/kg Pembrolizumab | 2

2. Secondary Outcome: Dose Limiting Toxicities (DLTs)
Description: Evaluate the DLTs of MK-3475 in combination with BCG in this population. DLTs will be defined as significant adverse events occurring during the DLT observation period (2 week pre-induction phase and the 7 weeks of induction phase) that is related to either drug or the combination. DLT will be evaluated according to CTCAE v 4.03 criteria.
Time Frame: Up to 9 weeks
Measure: Number; unit: DLT Event
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC)
Number analyzed (Participants) | 3 | 6
DLT Event | 0 | 1

3. Secondary Outcome: Incidence of Adverse Events
Description: Determine the safety and tolerability of the combination of MK-3475 and BCG in subjects with high risk or BCG-refractory non-muscle-invasive bladder cancer by evaluating the number, frequency, and severity of adverse events using CTCAE v 4.03. This table provides the number of patients with their worst grade toxicity for any AEs a patient experienced and AEs that were found to have a possible, probable, or definite attribution with at least one of the study treatment agents.
Time Frame: Up to 30 days from the last dose of study drug, up to 2.5 years
Measure: Number; unit: participants
Groups:
- Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC): PRE-INDUCTION PHASE: Patients receive pembrolizumab intravesically once on day -14.
  INDUCTION PHASE: Patients receive BCG solution intravesically once weekly for 6 weeks at weeks 0-5 and pembrolizumab intravesically every 2 weeks at weeks 0, 2, and 4.
  MAINTENANCE PHASE: Beginning 2 weeks after the last dose of BCG solution, patients receive pembrolizumab intravesically every 2 weeks for 12 weeks at weeks 7, 9, 11, 13, 15, and 17 for a total of 6 doses. Patients then receive pembrolizumab intravesically every 4 weeks at weeks 21, 25, 29, 33, 37, 41, 45, and 49 for a total of 8 doses.
  BCG Solution: Given intravesically Laboratory Biomarker Analysis: Correlative studies Pembrolizumab: Given intravesically Pharmacological Study: Correlative studies
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC)
Number analyzed (Participants) | 3 | 6
participants
  All Adverse Events Grades 1-2 | 0 | 3
  All Adverse Events Grade 3 | 3 | 2
  All Averse Events Grade 5 | 0 | 1
  Pembrolizumab Attributed Adverse Events Only Grade 1-2 | 3 | 4
  Pembrolizumab Attributed Adverse Events Only Grade 5 | 0 | 1
  BGC Attributed Adverse Events Only Grade 1-2 | 3 | 6

4. Other Pre Specified Outcome: Change in Cytokines in the Blood
Description: Blood will be collected for measurement of cytokines in order to explore humoral and cellular responses to MK-3475 and BCG treatments. Cytokines will be measured using ELISA assays.
Time Frame: At weeks -2, 0, and 17
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Change in Cytokines in Urine
Description: Urine will be collected for measurement of cytokines in order to explore humoral and cellular responses to MK-3475 and BCG treatments. Cytokines will be measured using ELISA assays.
Time Frame: Up to week 49
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Expression of PD-L1
Description: Expression of tumor biomarker PD-L1 as defined by immunohistochemistry (IHC) will be assessed and results will be correlated with adverse effects and recurrence rate. This evaluation will be performed on archived tissue samples obtained at baseline and on fresh tissue from any subsequent biopsies.
Time Frame: At baseline and then up to 49 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Expression of PD-1
Description: Expression of tumor biomarker PD-1 as defined by immunohistochemistry (IHC) will be assessed and results will be correlated with adverse effects and recurrence rate. This evaluation will be performed on archived tissue samples obtained at baseline and on fresh tissue from any subsequent biopsies.
Time Frame: At baseline and then up to 49 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Expression of PD-L2
Description: Expression of tumor biomarker PD-L2 and immune cell infiltration as defined by immunohistochemistry (IHC) will be assessed and results will be correlated with adverse effects and recurrence rate. This evaluation will be performed on archived tissue samples obtained at baseline and on fresh tissue from any subsequent biopsies.
Time Frame: At baseline and then up to 49 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Lymphocyte Profile
Description: Peripheral blood will be taken for evaluation of a lymphocyte profile which will be analyzed using automated flow cytometric techniques and will measure humoral and cellular response to tumor antigens.
Time Frame: At weeks -2, 0, and 17
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Plasma Concentration-time Profile
Description: Blood serum concentrations of MK-3475 will be evaluated during pre-induction (week -2) at baseline (0 minutes) and at 15, 30, and 60 minutes post-dosing for determination of plasma PK parameters.
Time Frame: Week -2: At minute 0, then 15, 30, and 60 minutes post-dosing
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Plasma Concentration-time Profile
Description: Blood serum concentrations of MK-3475 will be evaluated during induction (week 4) at baseline (0 minutes) and at 15, 30, and 60 minutes post-dosing for determination of plasma PK parameters.
Time Frame: Week 4: At minute 0, then 15, 30, and 60 minutes post-dosing
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Urine Concentration-time Profile
Description: Urine concentrations of MK-3475 will be evaluated during induction (week -2) at 30 minutes prior to dosing and 2 hours post-dosing for determination of urine concentration-time profile.
Time Frame: Week -2: At 30 minutes prior to dosing and 2 hours after dosing
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Urine Concentration-time Profile
Description: Urine concentrations of MK-3475 will be evaluated during induction (week 4) at 30 minutes prior to dosing and 2 hours post-dosing for determination of urine concentration-time profile.
Time Frame: Week 4: At 30 minutes prior to dosing and 2 hours after dosing
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Response Rate
Description: Determine the response rate in terms of complete pathologic response in this population will be assessed when the patient undergoes cystoscopies. Patients will be examined via bladder cystoscopy and may undergo biopsy for pathological confirmation if needed. Responses will be categorized as yes or no for bladder recurrence.
Time Frame: At baseline and up to 49 weeks
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Tumor Progression
Description: The progression rate of the tumor will be defined as positive transurethral resection and/or biopsy.
Time Frame: Up to 49 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were collected over a 3 year period. Each patient was followed from the time of treatment, during treatment at the beginning of each cycle through 30 days post last treatment.
Arm/Group | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC)
All-Cause Mortality (participants affected / at risk) | 1/3 | 3/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/6
Other Adverse Events (participants affected / at risk) | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) (N=3) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC) (N=6)
Myocardial Infarctrion (Cardiac disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Autoimmune Disorder (Immune system disorders) | 0 (0) | 1 (2)
Pelvic Infection (Infections and infestations) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I: Cohort 1 (1 mg/kg Pembrolizumab, 50 mg BGC) (N=3) | Phase I: Cohort 2 (2 mg/kg Pembrolizumab, 50 mg BGC) (N=6)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 3 (9) | 4 (5)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (5) | 0 (0)
Cardiac troponin I increased (Investigations) | 1 (1) | 0 (0)
Creatinine increased (Investigations) | 2 (10) | 5 (7)
Diarrhea (Gastrointestinal disorders) | 1 (2) | 3 (9)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 3 (6) | 6 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2) | 1 (1)
Hypertension (Vascular disorders) | 3 (24) | 6 (31)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (5) | 3 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 1 (2)
Proteinuria (Renal and urinary disorders) | 2 (4) | 5 (7)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2) | 2 (3)
Urine discoloration (Renal and urinary disorders) | 1 (3) | 1 (1)
Alkaline phosphatase increased (Investigations) | 0 (0) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 2 (11)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain during urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Dysuria: A disorder characterized by painful urination. (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary urgency (Renal and urinary disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-26): https://cdn.clinicaltrials.gov/large-docs/43/NCT02808143/Prot_SAP_000.pdf